CLINICAL TRIAL: NCT07363850
Title: A Study to Evaluate the Effectiveness of Group Gaming Interventions for Individuals With Problematic Gaming Behavior and Gaming Disorder.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NZhong-008
Record Dates: First submitted 2025-11-19; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-10

CONDITIONS: Gaming Disorder
Keywords: Gaming Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Behavioral: group gaming interventions
- control group (No Intervention)

INTERVENTIONS:
Behavioral: group gaming interventions — Each intervention is once a week for 90 minutes. A total of 10 sessions are set up, divided into the beginning stage (the 1st and the 2nd sessions), the middle stage (the 3rd to 8th), and the end stage (the 9th and 10th sessions). At this stage, the leader distributes point cards and wish lists to each member and explains the scoring rules, updating scores at the end of each activity. The point system combines group and individual scoring for cumulative totals. Each member may list desired prizes on their wish list, which will be redeemed for rewards based on their point total when the group concludes. The main aim of the middle stage is to knowledge game types, learn game reward mechanisms, the concept of IGD and influencing factors, and how to play healthily. In the end stage, each subgroup needs to show their complete game design, including the game name, game character, game rule, and reward mechanism, and all participants will make a summary of the whole process and say farewell
  Arms: intervention group

SUMMARY:
This is a randomized, parallel-group, two-arm study design registered with the Chinese Clinical Trial Registry. The study divides participants into an intervention group and a control group in the same ratio. The participants in the intervention group will receive a series of game-based activities and treatment. Firstly, we will distribute the recruitment advertisements for this intervention program in the school, including the project introduction, registration code, and contact details. Secondly, if students are interested in this project, they need to screen the code, and completely fill in personal information, and the screening questionnaire. Thirdly, students reaching the inclusion criteria and their parents will be invited to participate in a project briefing session and obtain their informed consent. Lastly, three times assessments in the whole process will be conducted, preintervention(T0), post-intervention(T1), and at a three-month(T3) follow-up. Importantly, participants can quit the project at any time during the whole process.

ELIGIBILITY:
Inclusion Criteria:

* (1) Clinical diagnosis of hazardous gaming defined in the ICD-11 (2) Fully comprehending the research's purpose and procedures and signing the informed consent

Exclusion Criteria:

* (1)Serious physical illness or intellectual disability (2) Clinical diagnosis of gaming disorder (3) Not completing all the interventions or assessments

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
the severity of gaming disorder | baseline, two months after intervention
  Description: Measured by Gaming Disorder Screening Scale

SECONDARY OUTCOMES:
average daily gaming hours | baseline, two months after intervention
  self-reported number of gaming sessions per week
frequency of gaming sessions | baseline, two months after intervention
  self-reported number of gaming sessions per week
anxiety severity | baseline, two months after intervention
  Measured by: Generalized Anxiety Disorder 7-item (GAD-7) Scale Scale Range: 0 to 21 (higher scores indicate worse anxiety)
depression severity | baseline, two months after intervention
  Measured by: Patient Health Questionnaire-9 (PHQ-9) Scale Range: 0 to 27 (higher scores indicate worse depression)
self-esteem | baseline, two months after intervention
  Measured by: Rosenberg Self-Esteem Scale (SES) Scale Range: 0 to 30 (higher scores indicate better self-esteem)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No